CLINICAL TRIAL: NCT00715962
Title: Efficacy and Safety of a Hospital Walking Program for Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E6326-W
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Acute Disease
Keywords: Hospitalization; Aged
MeSH Terms: conditions — Acute Disease | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobility Group (Active Comparator): The Walking Intervention includes assistance to walk twice daily with or without a rolling walker. In addition, a behavioral intervention that included goal setting and discussion of how to overcome mobility barriers was used to encourage the mobility group to be more active throughout hospital stay. Participants will keep a diary of out of bed activity and will be encouraged to set goals for additional out of bed activity daily.
  Interventions: Behavioral: Behavioral intervention; Other: Walking Intervention
- Control Group (Placebo Comparator): The control group will receive twice daily friendly visits to counter the attention being paid to the intervention group. They will complete a diary but of visitors to their room.
  Interventions: Other: Friendly visits

INTERVENTIONS:
Behavioral: Behavioral intervention — Using social cognitive theory, participants in the walking program group will be encouraged to complete a brief diary about out of bed activities like sitting up for meals of walks to the bathroom. They will be provided with information regarding the importance of being out of bed a praise for any attempts. They will be asked to set out of bed time activity goals daily. The control group will have a diary to track visitors.
  Arms: Mobility Group
Other: Walking Intervention — Participants in the walking program will be assisted to walk twice a day by trained staff. Those in the control group will be visited twice a day for friendly visits only
  Arms: Mobility Group
Other: Friendly visits — The control group will receive twice daily friendly visits and will be asked to complete a diary each day of the people who visit them in the hospital.
  Arms: Control Group

SUMMARY:
Low mobility, defined as being limited to bed or chair, is common during acute hospitalization. This study will evaluate the impact and safety of a hospital walking program for older patients during acute general medical hospitalization. Participants who are 65 years of age or older, will be randomized to usual care (UC) or to a hospital walking program (WP), which includes twice daily walks with assistance, provision of necessary ambulatory devices, and a behavioral intervention strategy designed to encourage out of bed activity. Throughout hospitalization, the WP and UC veterans will were wireless monitors on the thigh and ankle that measure activity. The primary goal will be in increase the length of time veterans spend out of bed and to assure this out of bed activity is safe.

DETAILED DESCRIPTION:
Background: Low mobility, defined as being limited to bed or chair, is common during acute hospitalization. The candidate's work has demonstrated low mobility to be associated with adverse outcomes including functional decline, need for new nursing home admission, and death even after controlling for illness severity and comorbidity. Objective: Using a Phase II trial design, the impact and safety of a hospital walking program for older patients during acute general medical hospitalization will be evaluated.

Project Design: 100 patients, age 65 years admitted to the medical wards at the Birmingham VAMC will be recruited within 48 hours of hospitalization and followed for 14 days after enrollment or until discharge, which ever comes first. Exclusion criteria will include: (1) Delirious based on positive Confusion Assessment Method (CAM); (2) Mini Mental State Examination Score < 17; (3) Patient on isolation; (4) Inability to ambulate 2 weeks prior to admission; (5) Having a medical diagnosis deemed by the primary physician to be a contraindication to ambulation; (6) patient with an imminently terminal illness; and (7) Non-English speaking. Participants will be randomized to either usual care (UC) or to a hospital walking program (WP), which includes twice daily walks with assistance, provision of necessary ambulatory devices, and a behavioral intervention strategy designed to encourage out of bed activity. Throughout hospitalization, the WP and UC veterans will wear on the ipsilateral thigh and ankle wireless monitors that measure horizontal and vertical orientation with respect to gravity. Previously validated by the candidate to assess levels of mobility during hospitalization, the output will be used to calculate the length of time patients spent lying, sitting, and standing or walking, using pre-defined criteria. Other daily measures will include orthostatic blood pressure, functional assessments, and assessment of falls and symptoms over the previous 24-hours. The primary outcome measure is time out of bed as measured by the wireless monitors. Importantly, our goal is to assess not only the amount of mobility that occurred as a result of the hospital walking program but that which occurred beyond the intervention. In our previous VA-funded study, patients spent an average of 17.1% or 4.1 hours out of bed per 24-hour period of time (s.d. 2.9). Our goal is to increase this by 50% or 2 hours to an average of 6.1 hours. This results in an effect size of 0.69 standard deviation units. A sample size of 45 per group provides 90% power to detect this 2-hour difference in the amount of time patients spend out of bed at the = .05 level.

Significance: at present there is a paucity of data regarding the impact or safety of a hospital walking program for general medical patients. Results of this study will enable researchers to determine the safety and efficacy of the walking program for older veterans during hospitalization and will provide information regarding effect size for a definitive intervention trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 65 years;
2. Admitted to the Birmingham VAMC for a medical condition

Exclusion Criteria:

1. Delirious based on positive Confusion Assessment Method (CAM);
2. Mini-Cognitive Assessment score indicating dementia;
3. Inability to ambulate 2 weeks prior to admission;
4. Having a medical diagnosis deemed by the primary physician to be a contraindication to ambulation;
5. patient with an imminently terminal illness; and
6. Non-English speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J. Brown, MD MSPH, Principal Investigator — VA Medical Center, Birmingham
Locations (1):
- VA Medical Center, Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Persons interested in obtaining the dataset will be asked to complete a data sharing agreement and procure IRB approval from their institution. At that time a de-identified dataset will be provided to them.

REFERENCES:
- [Derived] Brown CJ, Foley KT, Lowman JD Jr, MacLennan PA, Razjouyan J, Najafi B, Locher J, Allman RM. Comparison of Posthospitalization Function and Community Mobility in Hospital Mobility Program and Usual Care Patients: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jul 1;176(7):921-7. doi: 10.1001/jamainternmed.2016.1870. PMID 27243899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were patients 65 years or older admitted to the medical wards of the Birmingham Veterans Affairs Medical Center from January 12, 2010 to June 29, 2011.
Pre-assignment Details: Inclusion criteria were: having a negative screen for cognitive impairment (Mini Cog score ≥ 3), not being delirious (CAM score=0), self-report of being ambulatory with or without an assistive device in the 2 weeks before admission, not having a significant language barrier requiring a translator, and not previously enrolled in the study.
Groups:
- Mobility Group: Participants will receive assistance to walk twice daily, plus encouragement to be more active throughout hospital stay. Participants will keep a diary of out of bed activity and will be encouraged to set goals for additional out of bed activity daily.
  Behavioral encouragement of out of bed activity: Using social cognitive theory, participants in the walking program group will be encouraged to complete a brief diary about out of bed activities like sitting up for meals of walks to the bathroom. They will be provided with information regarding the importance of being out of bed a praise for any attempts. They will be asked to set out of bed time activity goals daily. The control group will have a diary to track visitors.
  Walking Intervention: Participants in the walking program will be assisted to walk twice a day by trained staff. Those in the control group will be visited twice a day for friendly visits only
- Control Group: The control group will receive twice daily friendly visits. They will complete a diary but of visitors to their room.
  Friendly visits: The control group will receive twice daily friendly visits and will be asked to complete a diary each day of the people who visit them in the hospital.
Period: Overall Study
Arm/Group | Mobility Group | Control Group
Started | 50 | 50
Completed | 44 | 48
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Population: Participants were 100 patients aged 65 years or older admitted to the medical wards of the Birmingham Veterans Affairs Medical Center (BVAMC).
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobility Group | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 50 | 50 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 48 | 49 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 39 | 42 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Mobility Knowledge PreTest Score [Mean (Standard Deviation); unit: units on a scale] — Scale range 0-5 with higher scores indicating higher knowledge regarding importance of mobility during hospitalization.
  units on a scale | 2.4 (1.1) | 2.6 (1.1) | 2.5 (1.1)
Falls Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — The participant was asked "On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all, how confident are you that you can do the following activities without falling?". Each item is scored from 1 to 10, and the responses are summed for all 10 questions. The Falls Self-efficacy scale scores range from 10 - 100 with higher scores indicating lower confidence in ability to perform 10 different activities without falling.
  units on a scale | 15.8 (6.5) | 15.8 (6.2) | 15.8 (6.3)
Activities of Daily Living (ADL) 2 Weeks prior to admission [Mean (Standard Deviation); unit: units on a scale] — At baseline, patients were asked to rate their level of independence with 6 activities of daily living (feeding, bathing, dressing, toileting, transferring, and walking) in the two weeks prior to their hospital admission. They were asked if they were independent (score =1), needed some assistance (score = 2) or required total assistance with the activity (score = 3). Scores for all 6 ADLs were summed with a range of 6-18 with higher scores indicating less independence with ADLs.
  units on a scale | 7.96 (1.5) | 8.0 (1.8) | 8.0 (1.6)
ADL on Admission [Mean (Standard Deviation); unit: units on a scale] — At baseline, patients were asked to rate their current level of independence with six activities of daily living (feeding, bathing, dressing, toileting, transferring, and walking). They were asked if they were independent (score =1), needed some assistance (score = 2) or required total assistance with the activity (score = 3). Scores for each of the 6 ADLs were summed; scores ranged from 6-18 with higher scores indicating less independence with ADLs.
  units on a scale | 8.8 (2.7) | 9.1 (2.9) | 8.9 (2.8)
Life-Space Assessment score [Mean (Standard Deviation); unit: units on a scale] — The UAB Study of Aging Life-Space Assessment (LSA) is a validated tool that measures mobility and function based on the distance which a person reports moving during the four weeks preceding the assessment. Scores range from 0 - 120 with higher scores reflecting higher levels of community mobility.
  units on a scale | 53.9 (29.4) | 51.5 (21.1) | 52.7 (25.5)
Mini-Nutritional Assessment score [Mean (Standard Deviation); unit: units on a scale] — The Mini-Nutritional Assessment (MNA) is a 6-item screening test of risk for malnutrition. Responses to the questions are summed to provide a score, with a range from 0-14.
  12-14 points: Normal nutritional status 8-11 points: At risk of malnutrition 0-7 points: Malnourished
  units on a scale | 9.4 (2.6) | 9.0 (2.3) | 9.2 (2.4)
Short Nutritional Assessment Questionnaire (SNAQ) score [Mean (Standard Deviation); unit: units on a scale] — This 4-item questionnaire is used to determine risk of weight loss. Each question is scored from 1-5 and the questions are summed to give a SNAQ score. Scores range from 4 - 20 and SNAQ scores of ≤14 indicate significant risk of at least 5 % weight loss within six months.
  units on a scale | 13.7 (3.4) | 13.5 (3.3) | 13.6 (3.3)
Gait speed [Mean (Standard Deviation); unit: meters per second] — If able to walk a short distance, patients were asked to perform a timed 10-foot (3 meter) walk. Two walks were done with the faster of the two times being utilized for analysis. Gait speeds of > or = to 1.0 meters/sec are considered normal; slower gait speeds are associated with increased risk of adverse outcomes including falls, ADL decline, nursing home placement and death.
  meters per second | 0.50 (0.26) | 0.51 (0.26) | 0.51 (0.26)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: units on a scale] — The Geriatric Depression Scale-short form is a 15-item questionnaire to screen for the presence of depression. Answers to the 15 "yes or no" questions are summed with scores of 6 or greater being identified as a positive screen for depression.
  units on a scale | 4.7 (3.2) | 5.0 (3.0) | 4.8 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Falls
Description: Patients were asked daily during hospitalization to self-report any falls
Time Frame: 18 months
Measure: Number; unit: participants
Groups:
- Mobility Group: Participants will receive assistance to walk twice daily, plus a behavioral intervention that encouragement to be more active throughout hospital stay. Participants will keep a diary of out of bed activity and will be encouraged to set goals for additional out of bed activity daily.
  Behavioral encouragement of out of bed activity: Using social cognitive theory, participants in the walking program group will be encouraged to complete a brief diary about out of bed activities like sitting up for meals of walks to the bathroom. They will be provided with information regarding the importance of being out of bed a praise for any attempts. They will be asked to set out of bed time activity goals daily. The control group will have a diary to track visitors.
  Walking Intervention: Participants in the walking program will be assisted to walk twice a day by trained staff. Those in the control group will be visited twice a day for friendly visits only
Arm/Group | Mobility Group | Control Group
Number analyzed (Participants) | 50 | 50
participants | 0 | 2
Statistical Analysis 1: Comparison: Mobility Group vs Control Group; Test type: Superiority or Other; p < .05, Fisher Exact; Fisher's exact test used as the rate of falling was low

2. Secondary Outcome: Life-Space Assessment Score
Description: The UAB Study of Aging Life-Space Assessment (LSA) is a validated tool that measures mobility and function based on the distance which a person reports moving during the four weeks preceding the assessment. Life-space "levels" range from within one's dwelling to beyond one's town. A life-space composite score is calculated based on life-space level, degree of independence in achieving each level, and the frequency of attaining each level. Scores range from 0 - 120 with higher scores indicating greater community mobility.
Time Frame: 4-6 weeks after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobility Group | Control Group
Number analyzed (Participants) | 50 | 50
units on a scale | 52.5 (29.0) | 41.6 (21.5)
Statistical Analysis 1: Comparison: Mobility Group vs Control Group; Test type: Superiority or Other; p < .05, ANCOVA

3. Primary Outcome: Amount of Time Spent Out of Bed as Measured by Wireless Accelerometers
Description: Throughout the hospital stay, both the WP and UC patient wore a triaxial accelerometer on the ipsilateral thigh and ankle. The patient's skin was assessed regularly to assure there is no evidence of irritation. The wireless monitors were used to quantify the amount of mobility that occurs daily for each patient with researchers being blinded to the outcome.
Time Frame: During hospital stay
Population: Only data from those recording days during which sensors were worn for at least 12 hours, defined as a valid day recording, were considered for final analysis. The average out of bed activity (standing or walking) duration over valid days of recording for each person was reported.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Mobility Group | Control Group
Number analyzed (Participants) | 28 | 36
minutes/day | 43.0 (12.8) | 44.7 (10.1)

ADVERSE EVENTS:
Time Frame: 18 months
Description: To assess the safety of the walking intervention both UC and WP patients will be asked daily about the occurrence of falls in the previous 24-hours.
Arm/Group | Mobility Group | Control Group
Serious Adverse Events (participants affected / at risk) | 8/50 | 8/50
Other Adverse Events (participants affected / at risk) | 5/50 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobility Group (N=50) | Control Group (N=50)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) — To address the small risk of skin irritation, a gauze was used between the skin and the device and check the device at least daily for placement and signs of erythema and the device was moved to the opposite limb daily.
In hospital Falls (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Patients self-reported on falls in the prior 24 hours
Readmission (Surgical and medical procedures) | 4 (4) | 5 (5) — Readmission to the hospital within 30 days of discharge
Death (Surgical and medical procedures) | 2 (2) | 1 (1)
ICU Transfer (Surgical and medical procedures) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobility Group (N=50) | Control Group (N=50)
Fall post-hospitalization (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) — Patients were asked to report on any falls that occurred after hospital discharge.

LIMITATIONS AND CAVEATS:
Study may not be generalizable as subjects mostly male and not demented or delirious. Study sample is small and needs to be replicated in a larger cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No